CLINICAL TRIAL: NCT01455454
Title: Evaluation of the Feasibility of Rotational Thromboelastrometry During Cardiopulmonary Bypass Using a Heparinase Modified ROTEM® Assay
Brief Title: Heparin's Influence on ROTEM® Analysis
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Other Study IDs: 123/10
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- coronary artery disease: patients undergoing coronary artery bypass grafting using cardiopulmonary bypass

SUMMARY:
Coagulopathy with transfusion requirements is frequent during cardiac surgery with cardiopulmonary Bypass. Rotational thromboelastrometry (ROTEM®) is a viscoelastic whole blood point of care test used to assess the patient's coagulation status.

The purpose of this study is to evaluate the feasibility of ROTEM® analysis in the presence of very high heparin concentrations as seen during cardiopulmonary bypass.

DETAILED DESCRIPTION:
The Society of Cardiothoracic surgeons suggest that 50% of patients undergoing cardiac surgery have a blood transfusion.

Several studies indicate an increase in morbidity and mortality related to blood transfusions.

Traditionally, the coagulation tests are performed in the hematology laboratory.

Rotational thromboelastrometry is a useful method of assessing perioperative coagulation function in patients undergoing cardiac surgery.

The presence of significant amounts of heparin in blood samples during cardiopulmonary bypass induces artifactual errors when thromboplastin is used as a reagent. For this reason, whole blood coagulation monitoring with ROTEM® has not been feasible during cardiopulmonary bypass with heparin anticoagulation. Recently recombinant thromboplastin has come available. It's stability is guaranteed by the manufacturer for plasmatic heparin concentrations up to 5UI/l .

Three of the available ROTEM®-tests are EXTEM (activation by recombinant thromboplastin), INTEM (activation by elagic acid) and HEPTEM. In the latter, heparinase, added to the INTEM reagent, eliminates heparin to reveal underlying coagulopathies.

The purpose of this study is to evaluate the feasibility of ROTEM® analysis in the presence of very high concentration of heparin and to evaluate whether heparinase could reverse heparin's effect on EXTEM and INTEM during cardiopulmonary bypass.

Arterial blood samples were drawn for analysis after induction of anesthesia (T0),10 minutes after the administration of heparin (T1), at unclamping of the aorta (T2) and after heparin reversal with protamine (T3). The following tests will be performed: EXTEM, INTEM, HEPTEM and a heparinase modified EXTEM. For the latter, recombinant thromboplatin instead of the elagic acid is used in the HEPTEM test. Heparin concentrations are measured at T1 and at the end of bypass (T2). HEPCON® was used for heparin management.

ELIGIBILITY:
Inclusion Criteria:

* Patients ungergoing coronary artery bypass grafting using cardiopulmonary bypass
* Patients from 18 to 85 years old.

Exclusion Criteria:

* Patients incapable to consent.
* Known coagulopathies or platelet dysfunction.
* Patients treated with antiplatelet drugs other than aspirin.
* Patients treated with anti vitamine K anticoagulants.
* Patients treated with heparin less than 6 hours prior to surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary artery bypass grafting using cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline ROTEM® measurements after the administration of heparin
  Baseline ROTEM® measurement will be compared to ROTEM® measurements after the administration of heparin, at the end of cardiopulmonary bypass and after the administration of protamine.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo E Marcucci, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Gronchi F, Perret A, Ferrari E, Marcucci CM, Fleche J, Crosset M, Schoettker P, Marcucci C. Validation of rotational thromboelastometry during cardiopulmonary bypass: A prospective, observational in-vivo study. Eur J Anaesthesiol. 2014 Feb;31(2):68-75. doi: 10.1097/EJA.0b013e328363171a. PMID 23867776